CLINICAL TRIAL: NCT02773342
Title: An Evaluation of Sequential Computed Tomography of the Chest in Management of Invasive Pulmonal Aspergillosis in Neutropenic Patients With Haematological Malignancies
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital of Cologne (Other)
Responsible Party: Principal Investigator, Prof. Dr. Oliver A. Cornely, University Hospital of Cologne, University Hospital of Cologne
Other Study IDs: CT_IPA_NEUT
Record Dates: First submitted 2013-05-06; First posted 2016-05-16 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Invasive Aspergillosis
Keywords: Invasive Pulmonal Aspergillosis; Neutropenic Patients; Haematological Malignancies; Chest Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Pathological findings in chest CT

SUMMARY:
The incidence of invasive pulmonary aspergillosis (IPA) is increasing in all parts of the world. Despite introduction of new antifungal agents for prophylaxis and treatment of IPA in the last decade, the outcome of patients with IPA is still unsatisfactory and needs improvement. Particularly, recent developments in diagnostic imaging, including introduction of high-resolution computed tomography (CT) into standard procedures, made a place for improvement of diagnosis of IPA.

Computed tomography of the chest is the optimal, recommended imaging procedure for diagnosis of pneumonia in febrile neutropenic patients and it is significantly superior to conventional chest X-ray. However, the method is associated with some difficulties mostly due to the broad spectrum of pathological findings in patients with IPA and their evolution over time. This has been described in retrospective studies on relatively small groups of patients. Prospective studies on larger populations are still missing, as well as studies on combination of different diagnostic modalities e.g. diagnostic imaging and microbiology.

We recently published the results of the clinical trial: "A Phase II Dose Escalation Study of Caspofungin in Patients with Invasive Aspergillosis" which used caspofungin doses of 70 to 200 mg daily for the first line treatment of IPA. The maximum tolerated dose was not reached, but response rates were impressive with complete plus partial responses accounting for 54.3% and overall mortality at 12-week follow-up as low as 28.3%. There was a tendency towards higher doses yielding higher response rates.

For the majority of these patients we obtained serial chest CT. So, for the first time a patient population is at hand, in which the kinetics of infiltrates over time can be described.

The main objective is to describe the pathological findings in chest CT performed sequentially in IPA patients while receiving effective antifungal therapy. The specific objectives are:

1. Characteristics of pathological findings in sequential chest CTs

   * To describe the pathological findings (e.g. halo sign, air crescent sign and air consolidation) in sequential high resolution computed tomogrphy (HRCT) examinations
   * To calculate the incidence of individual pathological findings in sequential CT examinations
   * To calculate a total volume of fungal infiltrates in sequential CT examinations
2. Correlation of pathological findings in sequential CT with corresponding white blood count (WBC) and absolute neutrophil count (ANC)

   * To correlate the appearance or disappearance of individual pathological findings with WBC and ANC
   * To correlate the volume of fungal infiltrates in sequential CT examinations with WBC and absolute neutrophil count
3. Correlation of pathological findings in sequential CT with the serum galactomannan index

   * To correlate the appearance or disappearance of individual pathological findings with the serum galactomannan index
   * To correlate the volume of fungal infiltrates in sequential HRCT examinations with the serum galactomannan index
4. Correlation of pathological findings in sequential HRCT with outcome of IFI

   * To correlate the appearance or disappearance of individual pathological findings with outcome of IFI
   * To correlate the volume of fungal infiltrates in sequential HRCT examinations with outcome of IFI

ELIGIBILITY:
Inclusion Criteria:

* At least two subsequent, evaluable CT examinations of the chest performed while on study

Exclusion Criteria:

* Diagnosis of underlying disease other than haematological malignancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Immunocompromised patients with proven or probable invasive aspergillosis received caspofungin once daily as an intravenous infusion
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2013-06; Primary Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Overall survival (%) | 48 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Cologne, Cologne, North Rhine-Westphalia, Germany